CLINICAL TRIAL: NCT04735835
Title: Personalized Responses to Dietary Composition Trial 3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zoe Global Limited (Other)
Collaborators: Massachusetts General Hospital (Other); Stanford University (Other); Harvard School of Public Health (HSPH) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PREDICT 3
Record Dates: First submitted 2021-01-13; First posted 2021-02-03 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Diabetes; Heart Diseases; Diet Habit; Diet Modification; Healthy; Obesity; Metabolism; Microbial Colonization
Keywords: Gut microbiome; Personalised nutrition; Machine learning; Postprandial metabolism; Metabolic health
MeSH Terms: conditions — Diabetes Mellitus; Heart Diseases; Feeding Behavior; Obesity; Communicable Diseases | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dietary Intervention (Experimental): Dietary intervention using standardized test meals after which the postprandial metabolic response is measured.
  Interventions: Other: Dietary Intervention

INTERVENTIONS:
Other: Dietary Intervention — To carry out a dietary intervention using standardized test meals, where the participant's postprandial response to the meal is measured and is used to predict their postprandial responses to other foods, along with input variables including metabolic profile, anthropometry, sleep and exercise.

SUMMARY:
The PREDICT 3 study will build on previous research in over 2,000 individuals to further refine machine learning models that predict individual responses to foods, with the aim of advancing precision nutrition science and individualized dietary advice. The study incorporates both standardized and controlled dietary intervention, for the purpose of testing postprandial responses to specific mixed meals, in addition to a free-living period with a dietary record for measuring responses to a large variety of meals consumed in a realistic context, where the role of external factors (e.g. exercise, sleep, time of day) on postprandial responses may be determined. For the first time this PREDICT study is built on top of a commercial product which will allow access to a much larger group of participants who are already collecting large amounts of data through digital and biochemical devices that can contribute to science.

DETAILED DESCRIPTION:
Choice of design: The study is a single arm mechanistic intervention study.

Study population: The subject must have enrolled in the commercial ZOE testing program in order to apply for participation in the PREDICT 3 research program.

Screening Assessment: The study eligibility criteria listed below closely match to the commercial eligibility criteria, which ZOE users consent to before enrolling in the commercial program.

Study duration: Each participant will take part in the study for 6-14 days.

Dietary intervention: The dietary intervention will be carried out on up to 6 days with the option to continue monitoring for a total study period of 14-days. On day one, participants will be asked to fit glucose monitor. Over the following consecutive days, each participant will be instructed to eat 2 standardized meals. Participants are free to eat whatever they wish at all other times. The standardized meals will be provided to all participants by the study team via post. The foods included as part of these meals will be foods that are commonly consumed and can be made from products sold in US supermarkets. Participants will be asked to consume the entire amount of food indicated for the standardized meals and to record any left-over food via a digital app for which training will be provided at the start of the study. Following completion of standardized meal period, participants are free to eat and drink whatever they wish and will be asked to track all meals, snacks and drinks on their digital app. Participants will also be advised not to change their physical activity patterns during the course of the study.

Regular contact will be made with the participants via phone, their app and text messages for the period of the intervention to encourage compliance and answer any queries.

Anthropometry: The participant will be instructed to report height and weight.

Dietary and Lifestyle: Participants will be asked to complete a baseline questionnaire online, as well as a diet history questionnaire with portion sizes about the month preceding their study period. They will be asked to record on a daily basis their dietary, activity, and psychological data (e.g. hunger) using a digital mobile phone app. Training in all apps and equipment will be given through written and online instructions and via communications with the study support staff.

Digital devices: Participants will be asked to record daily dietary and activity information using digital apps and lifestyle information will be monitored using a wearable device. The continuous glucose monitor (Freestyle Libre, CGM) provides continuous glucose profiles for up to 14 days. The CGM will be inserted on the back of the upper arm, one day before participants begin dietary intervention. This will measure subcutaneous interstitial fluid glucose concentrations every 5 minutes. The CGM will be removed at the end of the intervention period by the participant. A contact number will be made available to participants for any inquiries or if any problems arise. Data from the CGM will be downloaded, and glucose profiles will be evaluated on the basis of data collected.

Meal responses: As a product user, the participant will consume standardized meals an additional day to the study intervention.

Blood samples: As a product user, the participant will collect postprandial blood on 1 day using finger-prick blood sampling.

Stool sample: As a product user, the participant will collect a stool sample on 1 day.

Digital app: As product users, participants will be asked to download an app designed specifically for this study, which provides diet logging functionality similar to widely used existing apps such as MyFitnessPal.

Participants will be asked to record and monitor the following information via the digital app:

* All food and drink they consume, with serving sizes and photos
* Sleep and physical activity patterns, including exercise
* Hunger and alertness ratings
* Psychological feeling of energy and mood
* Prescription and over-the-counter drug consumption

The app will be available in versions for iOS operating systems. The app will synchronize remotely with backend database servers, over an encrypted and authenticated API, and will support offline operation for when patients wish to record an entry without network coverage. This continuous background synchronization means that it will not be necessary to explicitly download data from the phone at the end of the study.

Following the 2020 pandemic of COVID-19, participants are asked to use the COVID-19 Symptom Tracker app to record their physical health symptoms, or lack thereof, attributable to COVID-19, as well as demographic and other health information to track the spread of disease in real time, and to potentially reveal risk factors for infection and severe illness.

Subcohort: An opt-in follow-on study will be offered to participants to follow dietary guidance from the ZOE app based on their PREDICT 3 results. During the first 4 weeks, participants will be given dietary guidance to follow from the ZOE app. Thereafter, for a period of up to 12 months, participants will be asked to report on outcome measures at regular intervals (monthly). Outcome measures will be reported before, during and after the 4 week period and include weight, bristol stool chart, bowel habits, hunger, energy, adherence to dietary advice, and app usage. Participants (UK only) will collect additional stool samples at variable intervals.

The data will be used to test the efficacy of the ZOE dietary advice in promoting weight loss and improvement of overall health, and may be stratified by age, sex, BMI, adherence and/or motivation to take part in the PREDICT 3 study.

Food Frequency Questionnaire Validation: A food-frequency questionnaire (FFQ) developed using the most frequently logged foods within the ZOE app will be validated against a 4-day period of food logging in the app as well as the commonly used US-based DHQ3 FFQ (target enrollment; n=100).

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the commercial ZOE testing program
* Any sex
* Minimum 18 years of age (minimum 19 years of age in Alabama and Nebraska due to state laws)
* Body mass index (BMI) of greater than or equal to 16.5 kg/m2.
* Living in the continental US states, other than in New York (excluded from the ZOE testing product also as they are unable to access the dried blood spot service provided by Quest), or living in the UK
* Able and willing to comply with the study protocol and provide informed consent.
* Under care for chronic medical conditions (including eating disorders, type 1 diabetes, type 2 diabetes), and confirm they have checked with their primary care physician that this study is safe for them (US cohort only)

Exclusion Criteria:

* Cannot safely eat the pre-made test meals which contain standard US ingredients, e.g. due to allergy or recent gastrointestinal surgery, or are unwilling to consume these foods.
* Are pregnant.
* Have had a heart attack (myocardial infarction), stroke/transient ischemic attack (TIA), or major surgery in the last two months.
* Are unable to read and write in English, as the ZOE app is only available in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250000 (Estimated)
Dates: Start 2020-07-20 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Glucose | 6-14 days
  Measurement of blood glucose by continuous glucose monitor (mmol/L)
Gut microbiome species richness | 1 day
  Species count in fecal sample (as part of ZOE testing program)
Blood Lipids | 1 day
  Measurement of baseline and 6-h post-prandial triglycerides (mmol/L) by dried blood sample (as part of ZOE testing program)
Hunger and appetite assessment | 6-14 days
  Self-reported in-app question on energy levels (categorical) (as part of ZOE testing program)
Glucose and HbA1c | 2 days
  Measurement of baseline glucose (mmol/L) and HbA1c (%) by dried blood sample (as part of ZOE testing program)

SECONDARY OUTCOMES:
Dietary assessment | 6-14 days
  Weighed food log
Anthropometry | 1 day
  Weight (kg) (as part of ZOE testing program)
Anthropometry | 1 day
  Height (cm) (as part of ZOE testing program)
Dietary assessment | 1 month
  Diet history and portion size questionnaire about the preceding month (as part of ZOE testing program)
Bowel Type and Habit | 6-14 days
  Measurement by Bristol Stool Chart and Questionnaire (as part of ZOE testing program)
Perceived Energy Assessment | 6-14 days
  Self-reported in-app question on energy levels (categorical) (as part of ZOE testing program)
Covid-19 symptom assessment | 6 months
  Self-reported demographic and physical health symptoms, or lack thereof, reported on a daily basis (as part of ZOE testing program)

OTHER OUTCOMES:
Adherence (in sub-cohort) | Time Frame: 12 months: Baseline, Weekly (0 to 4 weeks), monthly (5 to 52 weeks)
  Self-reported in-app question on daily frequency of adherence (categorical)
Hunger (in sub-cohort) | Time Frame: 12 months: Baseline, Daily (0 to 4 weeks), monthly (5 to 52 weeks)
  Self-reported in-app question on hunger levels (categorical)
Weight (in sub-cohort) | Time Frame: 12 months: Baseline, Weekly (0 to 4 weeks), monthly (5 to 52 weeks)
  Body Weight (kg)
Bristol Stool Category (in sub-cohort) | Time Frame: 12 months: Baseline, Daily (0 to 4 weeks), monthly (5 to 52 weeks)
  Self-reported in-app Bristol Stool chart question (categorical)
Bowel Frequency (in sub-cohort) | Time Frame: 12 months: Baseline, Daily (0 to 4 weeks), monthly (5 to 52 weeks)
  Self-reported in-app question on bowel frequency
Energy (in sub-cohort) | Time Frame: 12 months: Baseline, Daily (0 to 4 weeks), monthly (5 to 52 weeks)
  Self-reported in-app question on energy levels (categorical)
Waist Circumference (in sub-cohort) | Time Frame: 12 months: Baseline, monthly (4 to 52 weeks)
  Self-reported in-app question on waist circumference
Hip Circumference (in sub-cohort) | Time Frame: 12 months: Baseline, monthly (4 to 52 weeks)
  Self-reported in-app question on hip circumference

CONTACTS AND LOCATIONS:
Overall Officials: Tim Spector, PhD, Principal Investigator — Zoe Global Limited
Locations (2):
- Zoe US Inc., Needham, Massachusetts, United States
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No